CLINICAL TRIAL: NCT01334632
Title: Comparison of Incidence of Brachial Plexus Injury After Rotator Cuff Repair With Continuous Interscalene Block Versus Patient Controlled Analgesia Morphine
Brief Title: Incidence of Brachial Plexus Injury After Rotator Cuff Repair With Continuous Interscalene Block
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Change of practice in the department (Nerve stimulation technique abandoned)
Sponsor: Centre Hospitalier Universitaire Vaudois (Other)
Responsible Party: Department of Anaesthesia, Centre Hospitalier Universitaire Vaudois and University of Lausanne
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: CHUV-74-10
Record Dates: First submitted 2011-04-11; First posted 2011-04-13 (Estimated); Last update posted 2014-03-20 (Estimated); Status verified 2011-04

CONDITIONS: Brachial Plexus Injury
Keywords: Electrophysiological study; Nerve block; Analgesia, patient-controlled; Shoulder surgery
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Continuous interscalene block (Active Comparator): Continuous interscalene block with bolus ropivacaine 0.5% and then continuous infusion of ropivacaine 0.2% 4 - 6 ml/h, associated with paracetamol and ibuprofen. Each group will contain 60 patients.
  Interventions: Procedure: Continuous interscalene block
- PCA morphine (Placebo Comparator): Patients with iv self-administration of morphine, associated with paracetamol and ibuprofen. Each group will contain 60 patients.
  Interventions: Procedure: PCA morphine

INTERVENTIONS:
Procedure: Continuous interscalene block — The continuous interscalene block will be performed with ultrasound 30 minutes before the intervention.
  Arms: Continuous interscalene block
Procedure: PCA morphine — Postoperative with iv self-administration of morphine
  Arms: PCA morphine

SUMMARY:
Brachial plexus injury after shoulder surgery with continuous interscalene block is 2.4% at 1 month and 0% at 6 months, but may be higher with a systematic postoperative neurological examination. Indeed, femoral neuropathy after anterior cruciate ligament reconstruction is 24% at 6 weeks in a cohort of 20 consecutive patients systematically screened with an electromyogram. Brachial plexus injury may be the consequence of the surgery (direct lesion by traction) or the continuous interscalene block. The goal of this study is to define the etiology of this postoperative neuropathy.

DETAILED DESCRIPTION:
Rotator cuff surgery is associated with moderate to severe postoperative pain. Among different analgesic strategies, continuous interscalene block is reported to be an efficient method, reducing opioid consumption and allowing rapid rehabilitation; however, patients may develop a transient neuropathy after surgery, which could have a significant impact on active patients. This study is designed to compare the incidence of brachial plexus injury in two groups of patients: one with a continuous interscalene block, and one with a patient control analgesia of morphine (self-iv administration of morphine). All patients will have a clinical neurological exam with a preoperative electromyogram in order to rule out a pre-existing neuropathy. Another clinical neurological exam with electromyogram will be performed between 4 and 6 postoperative weeks and, if pathological repeated at 6 months, 9 months and 12 months. The surgery will be done under general anesthesia for all patients.

ELIGIBILITY:
Inclusion Criteria:

* patients planned for rotator cuff repair
* ASA 1, 2 and 3
* age 16 years and more

Exclusion Criteria:

* peripheral neuropathy
* pre-existing brachial plexus injury
* diabetes mellitus
* alcoholism
* drug addiction

Ages: 16 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-04; Primary Completion 2013-03 (Estimated); Study Completion 2013-11 (Estimated)

PRIMARY OUTCOMES:
Incidence of brachial plexus injury | 6 weeks
  Clinical neurological exam (diminished or absent bicipital, tricipital reflex, or sensory loss on electromyoneurogram (axon loss ratio, Hoffmann reflex, compound muscle action potentials, any fibrillation potentials of the muscle at rest) at 6 weeks. A control will be done at 3 months, 6 months and 9 months if a neuropathy is diagnosed.

CONTACTS AND LOCATIONS:
Overall Officials: Eric Albrecht, MD, Principal Investigator — Department of Anesthesia, Centre Hospitalier Universitaire Vaudois and University of Lausanne
Locations (1):
- Department of Anesthesia, Centre Hospitalier Universitaire Vaudois and University of Lausanne, Lausanne, Canton of Vaud, Switzerland